CLINICAL TRIAL: NCT02787811
Title: Factors Affecting Success of IUI in Women With Unexplained Infertility
Brief Title: Predictors of Success of IUI in Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 149
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Assisted Reproductive Techniques
Keywords: IUI; Pregnancy rate; predictors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregnant (Active Comparator): women with positive serum beta HCG done 14 days after Intrauterine insemenation
  Interventions: Device: Intrauterine insemenation
- Nonpregnant (Active Comparator): women with negative serum beta HCG done 14 days after Intrauterine insemenation
  Interventions: Device: Intrauterine insemenation

INTERVENTIONS:
Device: Intrauterine insemenation — Semen preparation processing hen intrauterine transfer after 24 hours of HCG triggering of ovulation

SUMMARY:
Superovulation will be conducted with 100 mg of oral clomiphene citrate (Clomifene; Young Poong Pharmaceutical, Incheon, Korea) for 5 days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of human menopausal gonadotropin (hMG;Menogon; FerringPharamceutical Co, Germany). When more than 2 dominant follicles reached a diameter of 17 mm or the urinary specimen showed positive results for luteinizing hormone (LH) surge, 5000 IU of hCG (Pregnyl; Organon, Oss, the Netherlands) was injected intramuscularly.

DETAILED DESCRIPTION:
Superovulation will conducted with 100 mg of oral clomiphene citrate (Clomifene; Young Poong Pharmaceutical, Incheon, Korea) for 5 days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of human menopausal gonadotropin (hMG;Menogon; FerringPharamceutical Co, Germany). When more than 2 dominant follicles reached a diameter of 17 mm or the urinary specimen showed positive results for luteinizing hormone (LH) surge, 5000 IU of hCG (Pregnyl; Organon, Oss, the Netherlands) was injected intramuscularly. Successful pregnancy after IUI was confirmed by ultrasound as one or more visible gestational sacs in the uterine cavity.

ELIGIBILITY:
Inclusion Criteria:

* These patients had at least 1 tube patent
* there were no significant intrauterine or pelvic abnormalities demonstrated on pelvic-abdominal ultrasonography, hysteroscopy, and/or laparoscopy
* serum follicular stimulating hormone (FSH) level of12 mIU/mL or less

Exclusion Criteria:

* A woman's age of more than 40 years,
* ovarian cyst detected in the ultrasound examination
* uterine lesions such as submucosal leiomyoma, and a previous diagnosis of moderate to severe pelvic endometriosis.
* women with body mass index > 35 kg/m2,
* PCOS/anovulatory patients
* signs of hyperandrogenemia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
chemical pregnancy rate | 14 days after IUI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided